CLINICAL TRIAL: NCT04317586
Title: A Prospective, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Trident II Acetabular Shell in a Revision Indication
Brief Title: Trident II Revision Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79
Record Dates: First submitted 2020-03-12; First posted 2020-03-23 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Arthroplasty, Hip Revision
MeSH Terms: interventions — Second-Look Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Trident II Tritanium Acetabular Shell for Revision (Other)
  Interventions: Device: Trident II Tritanium Acetabular Shell for Revision

INTERVENTIONS:
Device: Trident II Tritanium Acetabular Shell for Revision — A hemispherical acetabular shell indicated for cementless application in a previously failed total hip arthroplasty (THA)

SUMMARY:
The purpose of this study is to review the performance and success rate of an FDA cleared cementless hip replacement part called the Trident II Tritanium Acetabular Shell. The study will specifically look at the need to revise the hip replacement after 5 years. This will be compared to how much this happens in patients who have hip replacement with similar cementless acetabular shells.

ELIGIBILITY:
Inclusion Criteria:

A. Patient has signed an IRB approved, study specific Informed Patient Consent Form.

B. Patient is a male or non-pregnant female age 18-85 years of age at the time of study device implantation.

C. Patient is a candidate for a revision of a failed acetabular component with a cementless acetabular component.

D. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations.

Exclusion Criteria:

E. Patient has a Body Mass Index (BMI) > 45. F. Patient is diagnosed with Inflammatory Arthritis. G. Patient has a non-Stryker retained stem. H. Patient has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.

I. Patient has a mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.

J. Patient has compromised bone stock which cannot provide adequate support and/or fixation to the prosthesis.

K. Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.

L. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days). M. Patient has a known sensitivity to device materials. N. Patient is a prisoner.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Lafayette General Orthopedic Center, Lafayette, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Beaumont Hospital Research Institute, Royal Oak, Michigan
  - The Orthopaedic & Fracture Clinic, P.A., Mankato, Minnesota
  - Reno Orthopedic Center Foundation, Reno, Nevada
  - OrthoNY, Albany, New York
  - Syracuse Orthopedic Specialists, New York, New York
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Hips Implanted
Period: Overall Study
Arm/Group | Trident II Tritanium Acetabular Shell for Revision
Started | 16; 17 Hips Implanted
Completed | 0; 0 Hips Implanted
Not Completed | 16; 17 Hips Implanted
Not completed — Participants/Hips Implanted Censored from Analysis | 2
Not completed — Participants Terminated Early (*15 Hips Implanted) | 14

BASELINE CHARACTERISTICS:
Population: 14 Participants, including one subject with bilateral hips implanted for a total of 15 Hips Implanted. All Demographic Data presented by Participant.
Units Other Than Participants: Hips Implanted
Arm/Group | Trident II Tritanium Acetabular Shell for Revision
Number analyzed (Participants) | 14
Number analyzed (Hips Implanted) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases Free From Trident II Acetabular Shell Revision
Description: To demonstrate, through absence of revision for aseptic loosening at five years postoperative, that acetabular revision with the Trident II Acetabular Shell provides clinical results comparable to similar acetabular components for revision indications. The study was terminated prior to the 5-year timepoint, data is presented through 2-years postoperative.
Time Frame: 6 Weeks, 3-6 Months, 1 Year and 2 Years
Population: One subject (1 Hip Implanted) did not return for a 6-Week Post-Operative Visit. Data are presented for 14 implanted for latest follow-up timepoint reached by each subject; presented at 6 Weeks (N=14 Hips Implanted), 3-6 Months (N=11 Hips Implanted), 1 Year (N=8 Hips Implanted) and 2 Years (N=2 Hips Implanted).
Measure: Count of Units; unit: Hips Implanted
Units Other Than Participants: Hips Implanted
Arm/Group | Trident II Tritanium Acetabular Shell for Revision
Number analyzed (Participants) | 13
Number analyzed (Hips Implanted) | 14
Hips Implanted
  Number of Hips Free From Revision at 6 Weeks | 14
  Number of Hips Free From Revision at 3-6 Months: number analyzed (Participants) | 10
  Number of Hips Free From Revision at 3-6 Months: number analyzed (Hips Implanted) | 11
  Number of Hips Free From Revision at 3-6 Months | 11
  Number of Hips Free From Revision at 1 Year: number analyzed (Participants) | 7
  Number of Hips Free From Revision at 1 Year: number analyzed (Hips Implanted) | 8
  Number of Hips Free From Revision at 1 Year | 8
  Number of Hips Free From Revision at 2 Years: number analyzed (Participants) | 2
  Number of Hips Free From Revision at 2 Years: number analyzed (Hips Implanted) | 2
  Number of Hips Free From Revision at 2 Years | 2

2. Secondary Outcome: Radiographic Stability
Description: Radiographic stability is a composite endpoint evaluating radiolucency and migration. Radiographic stability is defined as cases (hips implanted) which do not present with migration of greater than 5 mm in any direction or at least 2 mm radiolucency in all zones.
Time Frame: 6 Weeks and 3-6 Months
Population: Data reviewed by Independent Radiographic Reviewer is presented for one subject (1 Hip Implanted) at the 6 week and 3-6 Month timepoint. Following the initial review of 1 subject, the decision to terminate the study was made. No further radiographic review was conducted, and no additional radiographic stability data was collected.
Measure: Count of Units; unit: Hips Implanted
Units Other Than Participants: Hips Implanted
Arm/Group | Trident II Tritanium Acetabular Shell for Revision
Number analyzed (Participants) | 1
Number analyzed (Hips Implanted) | 1
Hips Implanted
  Hips Implanted that are Radiographically Stable at 6-Weeks | 1
  Hips Implanted that are Radiographically Stable at 3-6 Months | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from date of surgery to date of early termination, which was up to the 2 Year timepoint for the earliest enrolled subject.
Description: No difference of adverse event definition.
Arm/Group | Trident II Tritanium Acetabular Shell for Revision
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trident II Tritanium Acetabular Shell for Revision (N=14)
Deep Joint Infection (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitation: Early termination leading to small numbers of subjects analyzed due to lack of enrollment.

The Secondary Outcome of Radiographic Stability was corrected and adjusted to tabular presentation in alignment with the pre-specified endpoint in the study protocol, which is a composite endpoint of both Radiolucency and Migration. Radiographic Radiolucency as a standalone Secondary Outcome Measure was erroneously submitted in the original posting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT04317586/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT04317586/ICF_002.pdf